CLINICAL TRIAL: NCT01924208
Title: T Cell and Interferon Expression in Tonsils After Sublingual Immunotherapy and/or Nasal Live Attenuated Influenza Vaccine
Brief Title: Tonsillar Cytokine Expression After Allergen and/or Virus Intervention
Acronym: Tons2
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Turku University Hospital (Other Government)
Collaborators: Academy of Finland (Other); Juselius Foundation, Helsinki, Finland (Unknown); Foundation for Paediatric Research, Finland (Other); EVO special government transfers, Turku, Finland (Unknown)
Responsible Party: Principal Investigator, Tuomas Jartti, Dr, Turku University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Tons2
Record Dates: First submitted 2013-08-10; First posted 2013-08-16 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Healthy
Keywords: Timothy; Influenza; Interferon; T cell; Tonsil
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Timothy (Active Comparator): Allergen. Grazax® sublingual 75.000 SQ-T tablet (extracted from timothy, Phleum pretense), once daily until operation (ALK-Abelló, Hørsholm, Denmark) (n=30) .
  Interventions: Biological: Live attenuated influenza virus; Procedure: Timothy + attenuated influenza virus
- Live attenuated influenza virus (Active Comparator): Virus. Fluenz®, nasal live attenuated influenza vaccine, one 0.2 mL dose (MedImmune, Gaithersburg, USA) (n=60, 50:50 atopic:non-atopic).
  Interventions: Biological: Timothy, Phleum pretense; Procedure: Timothy + attenuated influenza virus
- Timothy + attenuated influenza virus (Active Comparator): Allergen. Grazax® sublingual 75.000 SQ-T tablet (extracted from timothy, Phleum pretense), once daily until operation (ALK-Abelló, Hørsholm, Denmark) + Virus. Fluenz®, nasal live attenuated influenza vaccine, one 0.2 mL dose (MedImmune, Gaithersburg, USA) (n=30).
  Interventions: Biological: Timothy, Phleum pretense; Biological: Live attenuated influenza virus
- No intervention (No Intervention): No intervention (n=60, 50:50 atopic:non-atopic).

INTERVENTIONS:
Biological: Timothy, Phleum pretense — Allergen. Grazax® sublingual 75.000 SQ-T tablet (extracted from timothy, Phleum pretense), once daily until operation (ALK-Abelló, Hørsholm, Denmark) (n=30) .
  Arms: Live attenuated influenza virus; Timothy + attenuated influenza virus
Biological: Live attenuated influenza virus — Virus. Fluenz®, nasal live attenuated influenza vaccine, one 0.2 mL dose (MedImmune, Gaithersburg, USA) (n=60, 50:50 atopic:non-atopic).
  Arms: Timothy; Timothy + attenuated influenza virus
Procedure: Timothy + attenuated influenza virus — Allergen. Grazax® sublingual 75.000 SQ-T tablet (extracted from timothy, Phleum pretense), once daily until operation (ALK-Abelló, Hørsholm, Denmark) + Virus. Fluenz®, nasal live attenuated influenza vaccine, one 0.2 mL dose (MedImmune, Gaithersburg, USA) (n=30).
  Arms: Live attenuated influenza virus; Timothy

SUMMARY:
Hypotheses

1. Immunotherapy induces tolerogenic effects to allergens in T cell regulation in tonsils.
2. Influenza vaccination induces a strong interferon response and decreases Th2 response in tonsils.
3. Influenza vaccination as an adjuvant on immunotherapy induces a better response to immunotherapy.

DETAILED DESCRIPTION:
Background: Tonsils are the primary nasopharyngeal lymphoid tissue and constitute the first contact point of the immune system to allergens and infectious agents. A peripheral T cell repertoire exists in tonsils, and tonsils have an active role for inducing and maintaining peripheral tolerance to allergens. Intralymphatic immunotherapy is a promising alternative for a subcutaneous or sublingual immunotherapy. More data is needed on the interaction between the peripheral (tonsillar) T cell response and specific allergen exposure and impact of respiratory virus infections on tolerance induction. Objective: To study the effects of sublingual grass pollen immunotherapy and/or nasal live attenuated influenza vaccine on tonsillar T cell and interferon (IFN) expression. In addition, we collect material on the investigation of role of tissues in immune tolerance and chronicity in allergic diseases.

Patients: Human tonsil samples will be obtained from less than 30-year-old routine tonsillectomy patients after sublingual grass immunotherapy (n=30), nasal live attenuated influenza vaccine (n=30 for atopic; and n=30 for non-atopic) and immunotherapy+influenza vaccine intervention (n=30). Controls without age limit or intervention (n=580) will also be recruited. Of these, age and atopy-matched controls will be selected as comparator groups for each intervention trial (n=30 for atopic; and n=30 for non-atopic). Control group will also be used for investigation of role of tissues in immune tolerance and chronicity in allergic diseases, immunomodulatory effects of respiratory viruses main focus being on human bocavirus and human rhinovirus infections, and in the search of new respiratory viruses.

Design: Study intervention products will be administered openly but the immunology outcomes will be analysed blindly.

Main outcomes: Gene expressions of IFN and T cell related genes will be the main outcomes and compared between intervention groups and correlated with the number of allergen extract doses or time from nasal influenza vaccination. Systemic immunologic outcomes (in peripheral blood mononuclear cells, blood RNA expression profiles, antibodies and cytokines in serum) will also be studied. The analyses include immunogenetics, virology, bacteriology and sensitization status. Clinical symptom scores will be recorded during the next 12 months from the screening visit.

Anticipated results: We expect that our tonsil approach will offer a new in vivo model for the understanding immune tolerance induction and will give new insights to the immunologic mechanisms in lymphoid tissue level. We hope to demonstrate that the immunologic effects of sublingual pollen immunotherapy can be modified with a nasal live attenuated influenza vaccine and thereby it should give basis for other add-on treatments aiming for more effective immunotherapy. The influenza virus vaccine is expected to promote Th1 cell expression over Th2 cell expression. Since the immunologic outcomes will be correlated to clinical efficacy during next influenza and pollen seasons, we hope to understand the clinical significance of the immunologic outcomes.

Innovation and impact: The unique strength of the project is to answer essential questions on development of allergen tolerance and a protective vaccine response in a human in vivo situation that cannot be answered in other settings. The proposed investigations may substantially enlarge our knowledge on the pathogenesis of organ directed allergic and non-allergic inflammation in humans, because the experiments will be performed directly with disease associated human cells and tissues. We expect that novel genes and pathways of immune regulation can be identified in tonsils by a detailed investigation of human immune response development to sublingual immunotherapy and influenza vaccine. The transcriptome and epigenome of these groups and further analyses of the role of T cells, B cells and innate lymphoid cells will provide essential information particularly on differences between atopic and non-atopic individuals, and anti-vaccine responses, natural viral infection, chronic viral infection, mechanisms of hypertrophic tonsillitis versus recurrent tonsillitis. The identification of new immune tolerance and immune activation pathways involved in the regulation of tissue cells is expected to provide novel knowledge for many other diseases in addition to asthma, because dysregulated immune system activation occurs in various human disorders such as cancer, autoimmunity, transplantation rejection and chronic infections.

ELIGIBILITY:
Inclusion Criteria:

* elective tonsillectomy with or without adenotomy according to clinical indication
* age >4 and <30 years
* written informed consent from the study subject or his/her guardian
* Fluenz® will be used for ages >4 and <30 years, i.e. off-label use of ages >18 and <30 years

Exclusion Criteria:

* systemic anti-inflammatory medication within prior 4 weeks
* systemic diseases affecting the immune system e.g. autoimmune diseases, immune complex diseases or immune deficiency diseases other than allergy, asthma or atopic dermatitis
* malignancy, depression, psychiatric illness or medication; planned vaccination during the study period (vaccinations should not be given during study period)
* forced expiratory volume in 1 second (FEV1) is under 80% of normal value or asthma is in a bad balance for those patients who would participate in the immunotherapy
* sublingual grass pollen will not be given for children under the age of 5
* additional exclusion criteria for Grazax® include hypersensitivity to any of the excipients (gelatin [fish source], mannitol, sodium hydroxide), inflammatory conditions in the oral cavity with severe symptoms such as oral lichen planus with ulcerations or severe oral mycosis, patients with uncontrolled or severe asthma (in adults: FEV1 < 70% of predicted value after adequate pharmacologic treatment, in children: FEV1 < 80% of predicted value after adequate pharmacologic treatment)
* addition exclusion criteria for Fluenz® include hypersensitivity to the active substances, to any of the excipients (sucrose, dibasic potassium phosphate, monobasic potassium phosphate, gelatin [porcine, Type A], arginine hydrochloride, monosodium glutamate monohydrate, gentamicin [a possible trace residue], eggs or to egg proteins [e.g. ovalbumin] and children and adolescents younger than 18 years of age receiving salicylate therapy because of the association of Reye's syndrome with salicylates and wild-type influenza infection

Ages: 4 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 180 (Estimated)
Dates: Start 2013-10; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Expressions of interferon and T cell and closely related cytokines and transcription factors in tonsils. | Up to 3 years
  Expressions of IFN-α, IFN-β, IFN-γ, IL-10, IL-13, IL-17, IL-28, IL-29, IL-37, TGF-β, FOXP3, GATA3, RORC2 and Tbet will be analyzed by quantitative real-time PCR.

CONTACTS AND LOCATIONS:
Overall Officials: Tuomas Jartti, M.D., Principal Investigator — Dept of Pediatrics, Turku University Hospital, Turku, Finland.; Cezmi Akdis, M.D., prof, Principal Investigator — Swiss Institute of Allergy and Asthma Research (SIAF), University of Zürich, Christine Kühne-Center for Allergy Research and Education (CK-CARE), Davos, Switzerland.
Locations (4):
- Finland (4):
  - Department of Otorhinolaryngology, Satakunta Central Hospital, Pori
  - Department of Otorhinolaryngology, Salo Regional Hospital, Salo
  - Department of Otorhinolaryngology, Turku University Hospital, Turku
  - Department of Pediatrics, Turku University Hospital, Turku

REFERENCES:
- [Background] Kucuksezer UC, Palomares O, Ruckert B, Jartti T, Puhakka T, Nandy A, Gemicioglu B, Fahrner HB, Jung A, Deniz G, Akdis CA, Akdis M. Triggering of specific Toll-like receptors and proinflammatory cytokines breaks allergen-specific T-cell tolerance in human tonsils and peripheral blood. J Allergy Clin Immunol. 2013 Mar;131(3):875-85. doi: 10.1016/j.jaci.2012.10.051. Epub 2012 Dec 23. PMID 23265862
- [Background] Palomares O, Ruckert B, Jartti T, Kucuksezer UC, Puhakka T, Gomez E, Fahrner HB, Speiser A, Jung A, Kwok WW, Kalogjera L, Akdis M, Akdis CA. Induction and maintenance of allergen-specific FOXP3+ Treg cells in human tonsils as potential first-line organs of oral tolerance. J Allergy Clin Immunol. 2012 Feb;129(2):510-20, 520.e1-9. doi: 10.1016/j.jaci.2011.09.031. Epub 2011 Nov 3. PMID 22051696